CLINICAL TRIAL: NCT06575088
Title: Effect of Cuff Pressure Level and Protective Padding Material Selection on the Prevention of Skin Complications in Pneumatic Tourniquet Applications in Upper Extremity Surgery: Clinical Research
Brief Title: Pneumatic Tourniquet Application in Upper Extremity Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, Sevgi Vermişli, Principal Investigator, Bursa City Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2022-12/5
Record Dates: First submitted 2024-08-22; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Skin Wound; Complication of Surgical Procedure
Keywords: Skin Complications; Protective Material; Pneumatic Tourniquet; Tourniquet Pressure; Upper Extremity Surgery

STUDY DESIGN:
Intervention Model Description: Patients were categorized into four groups based on the method of choice for determining the level of tourniquet cuff pressure and the PPM applied under the cuff. (i) . Standard tourniquet pressure (STP) with cotton pad; (ii) STP with elastic stockinette; (iii) limb occlusion pressure (LOP) with cotton pad; and finally, LOP with elastic stockinette. Power analysis was performed using the PASS software for sample size calculation. 50 patients were included in each group, considering that some patients might discontinue the trial. Block randomization method was used to randomize patients into study groups. The independent variables of the study were skin complications associated with tourniquet application on the skin under the sleeve. Complications were identified by the study team and confirmed by clinic nurses, and there was no disagreement regarding the occurrence of complications.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard tourniquet pressure with cotton pad (Active Comparator): Cotton pad was applied as protective filling material. Standard 250 mmHg pressure was applied as pneumatic tourniquet pressure.
  Interventions: Other: Standard tourniquet pressure (250 mmHg); Other: Cotton Pad
- Standard tourniquet pressure with elastic stockinette (Active Comparator): Elastic stockinette was applied as protective filling material. Standard 250 mmHg pressure was applied as pneumatic tourniquet pressure.
  Interventions: Other: Standard tourniquet pressure (250 mmHg); Other: Elastic stockinette
- Limb occlusion pressure with cotton pad (Active Comparator): Cotton pad was applied as protective filling material. Limb occlusion pressure was applied as pneumatic tourniquet pressure.
  Interventions: Other: Limb occlusion pressure; Other: Cotton Pad
- Limb occlusion pressure with elastic stockinette (Active Comparator): Elastic stockinette was applied as protective filling material. Limb occlusion pressure was applied as pneumatic tourniquet pressure.
  Interventions: Other: Limb occlusion pressure; Other: Elastic stockinette

INTERVENTIONS:
Other: Standard tourniquet pressure (250 mmHg) — The effectiveness of the protective padding material placed on the skin with a pneumatic tourniquet cuff and the pneumatic tourniquet pressure determination methods were compared.
  Arms: Standard tourniquet pressure with cotton pad; Standard tourniquet pressure with elastic stockinette
Other: Limb occlusion pressure — The effectiveness of the protective padding material placed on the skin with a pneumatic tourniquet cuff and the pneumatic tourniquet pressure determination methods were compared.
  Arms: Limb occlusion pressure with cotton pad; Limb occlusion pressure with elastic stockinette
Other: Cotton Pad — The effectiveness of the protective padding material placed on the skin with a pneumatic tourniquet cuff and the pneumatic tourniquet pressure determination methods were compared.
  Arms: Limb occlusion pressure with cotton pad; Standard tourniquet pressure with cotton pad
Other: Elastic stockinette — The effectiveness of the protective padding material placed on the skin with a pneumatic tourniquet cuff and the pneumatic tourniquet pressure determination methods were compared.
  Arms: Limb occlusion pressure with elastic stockinette; Standard tourniquet pressure with elastic stockinette

SUMMARY:
Purpose: This study investigated the effect of cuff pressure and the selection of protective padding material(PPM) on the prevention of skin complications associated with pneumatic tourniquet(PT) application in upper extremity surgery.

Methods: This randomized controlled trial was conducted between October 2022 and September 2023 at the Hand Surgery Clinic of XXX. Standard tourniquet pressure (STP) or limb occlusion pressure (LOP) was applied as PT cuff pressure. Cotton pads or elastic stockinette was used for PPM under the cuff. Patients were categorized into four groups; (i) STP with a cotton pad; (ii) STP with an elastic stockinette; (iii) LOP with a cotton pad; and (iv) LOP with an elastic stockinette. Total of 200 patients were included in the study, with 50 patients in each group. Skin complications were evaluated postoperatively at 0, 30, and 180 min.

DETAILED DESCRIPTION:
Pneumatic tourniquet (PT) is frequently used in extremity surgeries because of its advantages, including better surgical field visibility and shorter operation duration. Notwithstanding its advantages, PT can cause a number complications in the postoperative period, including pain, edema, skin complications, muscle injuries, thromboembolism, and neurological damage. Although the risks associated with the use of PT have decreased because of the introduction of adjustable pressure mechanisms and safety alarm systems, complications can still occur. Surgical team members should be knowledgeable about PT to ensure quality and safe patient care. It is of great importance to evaluate the size and shape of the extremity and skin condition prior to PT application, apply the appropriate size cuff, and evaluate the skin under the cuff and peripheral pulses distal to the cuff upon application.

There are different recommendations regarding safety practices for the application of PT in extremity surgeries. Previous studies in the relevant literature reported controversial results regarding the appropriate tourniquet cuff pressure for extremity surgery, and there are different applications for determining the cuff pressure. Previous studies mostly used standard tourniquet pressure (STP). STP is defined as 250 mmHg pressure for the upper extremity and 300 mmHg pressure for the lower extremity. Nevertheless, minimum inflation pressures have been recommended instead of STP to prevent complications likely associated with high pressures. Another method is the use of limb occlusion pressure (LOP). LOP is defined as the minimum pressure required to stop arterial blood flow into the extremity distal to the cuff. LOP can be determined manually or automatically by slowly inflating the cuff and stopping the pulse using certain equipment, including a Doppler flowmeter or pulse oximeter. It was suggested that PT cuff pressure could be minimized by LOP application and that the risk of tourniquet-related complications could be reduced. Most previous studies on PT have focused on the lower extremities. Nevertheless, tourniquet use also been the method of choice in upper extremity surgery to provide a surgical field without blood.

In PT applications, protective padding material (PPM) is placed between the skin and the cuff to prevent skin injuries. The Association of Perioperative Registered Nurses recommends the application of soft, low-lint padding materials, including limb protection sleeves or two layers of stockinette (plaster stocking). The padding material should not compress the skin or cause wrinkles. Fewer skin complications were observed in patients with cotton pads or elastic stockinette than in patients without PPM. There is no material with proven superiority in the use of PPM.

This study investigated the effects of cuff pressure level and the choice of PPM on the prevention of skin complications after PT in upper extremity surgery. It was hypothesized that there was a relationship between the level of cuff pressure and the PPM during use and skin complications during PT applications in upper extremity surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who 18 years and older
* Patients who undergoing upper extremity surgery
* Patients who underwent surgery under general and regional anesthesia
* Patients who having no communication problems
* Patients who agreeing to participate in the study

Exclusion Criteria:

* Patients who with communication barriers
* Patients who refused to participate in the study
* Patients who aged below 18 years
* Patients who underwent surgery for the second time
* Patients who underwent bilateral extremity surgery
* Patients without pneumatic tourniquet application
* Patients who received hypertension treatment
* Patients who diabetes mellitus treatment
* Patients who had skin lesions under the cuff during preoperative observation
* Patients who had active infection
* Patients who had skin complications
* Patients who have an above-elbow splint applied
* Patients who underwent surgical operation associated with malignancy
* Patients with the surgical area located proximal to the elbow

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Actual)
Dates: Start 2022-10-14 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Redness | through study completion, an average of 1 year
  Redness was defined as a reddish appearance on the skin, in contrast to a normal skin appearance.
Tourniquet scar | through study completion, an average of 1 year
  A tourniquet scar is a scar on the skin in the form of wrinkles and folds aligned with the structure of the sleeve.
Petechiae | through study completion, an average of 1 year
  Petechiae was defined as the occurrence of pinpoint-sized hemorrhages under the skin of the sleeve.
Bulla | through study completion, an average of 1 year
  A bulla is considered a fluid-filled blister on the skin.

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi Vermisli Ciftci, Ph.D., Study Chair — Republic of Turkey Ministry of Health Bursa City Hospital/Operating Room; Zeki Gunsoy, M.D., Principal Investigator — Republic of Turkey Ministry of Health Bursa City Hospital/Hand Surgery Clinic; Fatma Demir Korkmaz, Professor, Principal Investigator — Ege University/ Faculty of Nursing
Locations (1):
- Republic of Turkey Ministry of Health Bursa City Hospital, Bursa, Turkey (Türkiye)

REFERENCES:
- [Background] Aydin A, Kanan N. Effect of Protective Padding in Pneumatic Tourniquet Applications on the Prevention of Skin Complications. Orthop Nurs. 2022 Jul-Aug 01;41(4):260-268. doi: 10.1097/NOR.0000000000000857. PMID 35869912
- [Background] Jensen J, Hicks RW, Labovitz J. Understanding and Optimizing Tourniquet Use During Extremity Surgery. AORN J. 2019 Feb;109(2):171-182. doi: 10.1002/aorn.12579. PMID 30694553
- [Background] Bosman HA, Robinson AH. Pneumatic tourniquet use in foot and ankle surgery--is padding necessary? Foot (Edinb). 2014 Jun;24(2):72-4. doi: 10.1016/j.foot.2014.03.007. Epub 2014 Mar 25. PMID 24745802
- [Background] Din R, Geddes T. Skin protection beneath the tourniquet. A prospective randomized trial. ANZ J Surg. 2004 Sep;74(9):721-2. doi: 10.1111/j.1445-1433.2004.03143.x. PMID 15379794
- [Background] McMillan TE, Johnstone AJ. Tourniquet uses and precautions. Surg (United Kingdom). 2017;35(4):201-203. doi:10.1016/j.mpsur.2017.01.011
- [Background] Olivecrona C, Tidermark J, Hamberg P, Ponzer S, Cederfjall C. Skin protection underneath the pneumatic tourniquet during total knee arthroplasty: a randomized controlled trial of 92 patients. Acta Orthop. 2006 Jun;77(3):519-23. doi: 10.1080/17453670610012539. PMID 16819695
- [Background] Spruce L. Back to Basics: Pneumatic Tourniquet Use. AORN J. 2017 Sep;106(3):219-226. doi: 10.1016/j.aorn.2017.07.003. PMID 28865632
- [Background] Sun C, Yang X, Zhang X, Ma Q, Yu P, Cai X, Zhou Y. Personalized tourniquet pressure may be a better choice than uniform tourniquet pressure during total knee arthroplasty: A PRISMA-compliant systematic review and meta-analysis of randomized-controlled trials. Medicine (Baltimore). 2022 Feb 25;101(8):e28981. doi: 10.1097/MD.0000000000028981. PMID 35212310
- [Background] Martinez-Rico S, Lizaur-Utrilla A, Sebastia-Forcada E, Vizcaya-Moreno MF, de Juan-Herrero J. The Impact of a Phone Assistance Nursing Program on Adherence to Home Exercises and Final Outcomes in Patients Who Underwent Shoulder Instability Surgery: A Randomized Controlled Study. Orthop Nurs. 2018 Nov/Dec;37(6):372-378. doi: 10.1097/NOR.0000000000000501. PMID 30451774
- [Background] Bowen BA. Orthopedic Surgery. In: ROTHROCK JC, McEwen DR, eds. Alexander's Care of the Patient in Surgery. 16th ed. Optum/UnitedHealthCare San Antonio, Texas: Elsevier; 2018:2050-2300.
- [Background] Hicks RW, Denholm B. Implementing AORN recommended practices for care of patients undergoing pneumatic tourniquet-assisted procedures. AORN J. 2013 Oct;98(4):383-93; quiz 394-6. doi: 10.1016/j.aorn.2013.08.004. PMID 24075334
- [Background] Yalcinkaya M, Sokucu S, Erdogan S, Kabukcuoglu YS. Tourniquet use in orthopedic surgery: a descriptive survey study among Turkish orthopedic surgeons and residents in Istanbul. Acta Orthop Traumatol Turc. 2014;48(5):483-90. doi: 10.3944/AOTT.2014.14.0068. PMID 25429571
- [Background] Olaiya OR, Alagabi AM, Mbuagbaw L, McRae MH. Carpal Tunnel Release without a Tourniquet: A Systematic Review and Meta-Analysis. Plast Reconstr Surg. 2020 Mar;145(3):737-744. doi: 10.1097/PRS.0000000000006549. PMID 32097317
- [Background] Pinto A, Moniz J, Dinis A, Santos N, Carmona C. Pneumatic tourniquet in orthopedic surgery, an institutional good practices review. Reg Anesth Pain Med. 2022;47(Suppl 1):A1-A315. doi:10.1136/rapm-2022-ESRA.252 Background
- [Background] McEwen JA, Kelly DL, Jardanowski T, Inkpen K. Tourniquet safety in lower leg applications. Orthop Nurs. 2002 Sep-Oct;21(5):55-62. doi: 10.1097/00006416-200209000-00009. PMID 12432700
- [Background] Othman S, Pistorio AL, Lopez S, Orengia A, Born MW. Optimizing Tourniquet Pressure in Upper Extremity Surgery. J Hand Surg Asian Pac Vol. 2021 Dec;26(4):654-659. doi: 10.1142/S2424835521500636. PMID 34789106
- [Background] Morehouse H, Goble HM, Lambert BS, Cole J, Holderread BM, Le JT, Siff T, McCulloch PC, Liberman SR. Limb Occlusion Pressure Versus Standard Pneumatic Tourniquet Pressure in Open Carpal Tunnel Surgery - A Randomized Trial. Cureus. 2021 Dec 2;13(12):e20110. doi: 10.7759/cureus.20110. eCollection 2021 Dec. PMID 35003958
- [Background] Liu HY, Guo JY, Zhang ZB, Li KY, Wang WD. Development of adaptive pneumatic tourniquet systems based on minimal inflation pressure for upper limb surgeries. Biomed Eng Online. 2013 Sep 23;12:92. doi: 10.1186/1475-925X-12-92. PMID 24053348
- [Background] Drolet BC, Okhah Z, Phillips BZ, Christian BP, Akelman E, Katarincic J, Schmidt ST. Evidence for safe tourniquet use in 500 consecutive upper extremity procedures. Hand (N Y). 2014 Dec;9(4):494-8. doi: 10.1007/s11552-014-9667-1. PMID 25414611
- [Background] AORN Recommended Practices Committee. Recommended practices for the use of the pneumatic tourniquet in the perioperative practice setting. AORN J. 2007 Oct;86(4):640-655. doi: 10.1016/j.aorn.2007.09.004. No abstract available. PMID 18268836
- [Background] Hughes L, McEwen J. Investigation of clinically acceptable agreement between two methods of automatic measurement of limb occlusion pressure: a randomised trial. BMC Biomed Eng. 2021 May 8;3(1):8. doi: 10.1186/s42490-021-00053-9. PMID 33964963
- [Background] Tuncali B, Kokten G, Boya H, Altinel F, Kayhan Z. Efficacy of arterial occlusion pressure estimation-based tourniquet pressure settings in upper limb surgery. J Orthop Sci. 2022 Sep;27(5):1051-1055. doi: 10.1016/j.jos.2021.06.011. Epub 2021 Jul 24. PMID 34315653
- [Background] Masri BA, Day B, Younger AS, Jeyasurya J. Technique for Measuring Limb Occlusion Pressure that Facilitates Personalized Tourniquet Systems: A Randomized Trial. J Med Biol Eng. 2016;36(5):644-650. doi: 10.1007/s40846-016-0173-5. Epub 2016 Oct 4. PMID 27853415
- [Background] de Souza Leao MG, Neta GP, Coutinho LI, da Silva TM, Ferreira YM, Dias WR. Comparative analysis of pain in patients who underwent total knee replacement regarding the tourniquet pressure. Rev Bras Ortop. 2016 Sep 22;51(6):672-679. doi: 10.1016/j.rboe.2016.09.005. eCollection 2016 Nov-Dec. PMID 28050539
- [Background] Azad A, Sager B, Gupta S, Ayalon O, Paksima N. Reducing Tourniquet Pressures in Hand Surgery: Are Lower Pressures as Effective? J Wrist Surg. 2022 Sep 26;12(3):205-210. doi: 10.1055/s-0042-1753543. eCollection 2023 Jun. PMID 37223384
- [Background] Ishii Y, Matsuda Y. Effect of tourniquet pressure on perioperative blood loss associated with cementless total knee arthroplasty: a prospective, randomized study. J Arthroplasty. 2005 Apr;20(3):325-30. doi: 10.1016/j.arth.2004.10.001. PMID 15809950
- [Background] Unver B, Karatosun V, Tuncali B. Effects of tourniquet pressure on rehabilitation outcomes in patients undergoing total knee arthroplasty. Orthop Nurs. 2013 Jul-Aug;32(4):217-22. doi: 10.1097/NOR.0b013e31829aef2a. PMID 23881019
- [Background] Wu J, Fu Q, Li H, Han Y, Deng J, Chen Y, Qian Q. An alternative method for personalized tourniquet pressure in total knee arthroplasty: a prospective randomized and controlled study. Sci Rep. 2022 Jun 10;12(1):9652. doi: 10.1038/s41598-022-13672-6. PMID 35688920
- [Background] Kim TK, Bamne AB, Sim JA, Park JH, Na YG. Is lower tourniquet pressure during total knee arthroplasty effective? A prospective randomized controlled trial. BMC Musculoskelet Disord. 2019 Jun 4;20(1):275. doi: 10.1186/s12891-019-2636-7. PMID 31159799
- [Background] Oragui E, Parsons A, White T, Longo UG, Khan WS. Tourniquet use in upper limb surgery. Hand (N Y). 2011 Jun;6(2):165-73. doi: 10.1007/s11552-010-9312-6. Epub 2010 Dec 8. PMID 22654699
- [Background] Sato J, Ishii Y, Noguchi H, Takeda M. Safety and efficacy of a new tourniquet system. BMC Surg. 2012 Aug 15;12:17. doi: 10.1186/1471-2482-12-17. PMID 22894765
- [Background] Ekwunife RT, Iyidobi EC, Enweani UM, et al. Assessment of complications following use of pneumatic tourniquet for elective orthopedic procedures at National Orthopedic Hospital, Enugu. Int J Res Orthop. 2019;5(5):764. doi:10.18203/issn.2455-4510.intjresorthop20193822